CLINICAL TRIAL: NCT03529513
Title: Medibio Depression Diagnostic Aid Confirmatory Performance Study
Brief Title: Medibio DDA Confirmatory Performance Study
Status: Completed | Type: Observational
Sponsor: Medibio Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: MB-DEPDX04
Record Dates: First submitted 2018-01-29; First posted 2018-05-18 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Major Depressive Episode

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Depressed: Subjects currently experiencing a moderate-to-severe major depressive episode are clinically evaluated over approximately 2-week period. 24-hour ECG data recordings are collected during each of the two weeks. Subjects may continue on current treatment regimen.
  Interventions: Diagnostic Test: Medibio Depression Diagnostic Aid; Diagnostic Test: Mini International Neuropsychiatric Interview; Diagnostic Test: Hamilton Rating Scale for Depression - 17 Item
- Control: Subjects not currently experiencing a major depressive episode are clinically evaluated over approximately 2-week period. 24-hour ECG data recordings are collected during each of the two weeks. Subjects may continue on current treatment regimen.
  Interventions: Diagnostic Test: Medibio Depression Diagnostic Aid; Diagnostic Test: Mini International Neuropsychiatric Interview; Diagnostic Test: Hamilton Rating Scale for Depression - 17 Item

INTERVENTIONS:
Diagnostic Test: Medibio Depression Diagnostic Aid — The Medibio DDA processes the heart rate and actigraphy data from the third-party devices, characterizes these data in comparison to the benchmark patterns of persons currently experiencing a depressive episode.
Diagnostic Test: Mini International Neuropsychiatric Interview — The Mini International Neuropsychiatric Interview (M.I.N.I.) is a structured diagnostic interview that was developed as a simple tool to assist clinicians to conduct psychiatric diagnoses according to the DSM-IV and International Statistical Classification of Diseases and Related Health Problems tenth revision (ICD-10) criteria.
  Other Names: M.I.N.I.
Diagnostic Test: Hamilton Rating Scale for Depression - 17 Item — The clinician-administered Hamilton Depression Rating Scale (also known as the HAM-D) is the most widely used depression assessment scale . The original version contains 17 items (HDRS17) pertaining to symptoms of depression experienced over the past week. There are numerous versions with varying lengths that include the HDRS21, HDRS24, and HDRS29. This study will utilize the HDRS17 (HAMD-17) version.
  Other Names: HAMD-17

SUMMARY:
This study will determine whether the Medibio Depression Diagnostic Aid exceeds minimally acceptable thresholds for sensitivity and sensitivity in cases with a current depression episode and non-depressed controls.

DETAILED DESCRIPTION:
Subjects meeting study criteria will be enrolled into one of two study cohorts: a) outpatient individuals with current, moderate-to-severe major depressive episode (experimental group) and b) individuals without current major depressive episode that have been matched at the group level for age and gender (control group).

All subjects will undergo two separate psychiatric interviews to confirm current depression episode presence or absence. Thereafter subjects will wear a heart rate monitor on the chest to capture data over the course of 72 hours. Subjects will return approximately 1 week after initial placement of the monitor for equipment return and a safety check. Subjects will wear a heart-rate monitor over the course of 72 hours. Subjects will return within a week from the last visit for equipment return.

ELIGIBILITY:
All Subjects:

Inclusion Criteria:

* Subject is willing and able to provide consent.
* Subject has ability to read and understand the instructions for the study.
* Subject is willing to adhere to study procedures.

Exclusion Criteria:

* Subject has active psychotic symptoms.
* Subject has bipolar disorder.
* Subject has known, or is suspected to have a personality disorder.
* Subject has current suicidality of medium or high risk as determined by M.I.N.I. or HAMD-17 item #3 score of 3 of higher.
* Subject has history of central or obstructive sleep apnea OR STOP-BANG questionnaire score of ≥5.
* Subject has a pacemaker.
* Subject currently uses benzodiazepines on a scheduled basis.
* Subject currently uses chronotropic medication, such as beta-blockers, digoxin, sinoatrial/atrioventricular nodal-acting calcium channel blockers, or amiodarone.
* Subject is suspected or known to have active alcohol or drug abuse (including but not limited to abuse of marijuana).
* Subject has a terminal illness.
* For female subjects, subject is currently known to be pregnant or lactating.
* Subject has any other acute or chronic condition that in the investigators opinion would preclude the subject from being able to meet all of the protocol requirements, or would compromise the subject's safety during participation in the study, as judged by the investigator.
* Subject is currently participating in another clinical study. Subject currently uses antipsychotic medication for any indication.

Depressed Cohort Inclusion Criteria: Subject has current moderate or severe Major Depressive Disorder Episode, based on DSM-IV criteria for diagnosis as documented by clinician administered M.I.N.I plus HAMD-17 rating scale score ≥17.

Exclusion Criteria: Subject has presence of no or mild Major Depressive Disorder Episode, based on DSM-IV criteria for diagnosis as documented by clinician administered M.I.N.I OR HAMD-17 rating scale score <17.

Control Cohort Inclusion Criteria: Subject has no presence of mild, moderate, or severe Major Depressive Disorder Episode, based on DSM-IV criteria for diagnosis as documented by clinician administered M.I.N.I AND HAMD-17 rating scale score ≤7.

Exclusion Criteria: Subject has presence of mild, moderate, or severe Major Depressive Disorder Episode, based on DSM-IV criteria for diagnosis as documented by clinician administered M.I.N.I OR HAMD-17 rating scale score >7.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who may be currently experiencing an episode of depression that are being diagnosed or treated in a mental health setting.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Measure heart rate variability | Up to 2 weeks
  The Medibio Algorithm will process data from subject 24-hour ECG data recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Bruner, Study Director — Medibio Limited
Locations (8):
- United States (6):
  - CNS Network, Garden Grove, California
  - CNS Network, Torrance, California
  - Lindner Center of HOPE, Mason, Ohio
  - OCCI, Inc., Salem, Oregon
  - FutureSearch Trials, Dallas, Texas
  - White River Junction Veterans Affairs Medical Center, White River Junction, Vermont
- Australia (2):
  - Epworth Clinic, Camberwell, Victoria
  - The Melbourne Clinic, Richmond, Victoria

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.